CLINICAL TRIAL: NCT03677908
Title: Plasticity of Neonatal Neuronal Networks in Very Premature Infants: Source Localization of Temporal Theta Activity, the First Endogenous Neural Biomarker, in Temporoparietal Areas
Brief Title: Plasticity of Neonatal Neuronal Networks Temporal Theta Activity, the First Endogenous
Acronym: NEURONAUX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0048
Record Dates: First submitted 2018-09-14; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Premature Birth
Keywords: Temporoparietal Areas; Neural Biomarker
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 13 high: High-Density ElectroEncephaloGraphy analysis of 13 healthy premature infants
  Interventions: Other: ElectroEncephaloGraphy
- 15 low: Low-Density ElectroEncephaloGraphy analysis of other 15 healthy premature infants
  Interventions: Other: ElectroEncephaloGraphy

INTERVENTIONS:
Other: ElectroEncephaloGraphy — Density ElectroEncephaloGraphy analysis

SUMMARY:
Temporal theta slow-wave activity (TTA-SW) in premature infants is a specific signature of the early development of temporal networks, as it is observed at the turning point between non-sensory driven spontaneous local processing and cortical network functioning. The role in development and the precise location of TTA-SW remain unknown. Previous studies have demonstrated that preterms from 28 weeks of gestational age (wGA) are able to discriminate phonemes and voice, supporting the idea of a prior genetic structural or activity-dependent fingerprint that would prepare the auditory network to compute auditory information at the onset of thalamocortical connectivity. They recorded TTA-SW in 26-32 wGA preterms. The rate of TTA-SW in response to click stimuli was evalu- ated using low-density EEG in 30 preterms. The sources of TTA-SW were localized by high-density EEG using different tissues conductivities, head models and mathematical models.

DETAILED DESCRIPTION:
Temporal theta slow-wave activity (TTA-SW) in premature infants is a specific signature of the early development of temporal networks, as it is observed at the turning point between non-sensory driven spontaneous local processing and cortical network functioning. The role in development and the precise location of TTA-SW remain unknown. Previous studies have demonstrated that preterms from 28 weeks of gestational age (wGA) are able to discriminate phonemes and voice, supporting the idea of a prior genetic structural or activity-dependent fingerprint that would prepare the auditory network to compute auditory information at the onset of thalamocortical connectivity. They recorded TTA-SW in 26-32 wGA preterms. The rate of TTA-SW in response to click stimuli was evalu- ated using low-density EEG in 30 preterms.

ELIGIBILITY:
Inclusion Criteria:

* healthy premature infants
* Gestational Ages of 26 and 32 wGA

Exclusion Criteria:

* unhealthy premature infants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 28 healthy premature infants follow-up between the Gestational Ages of 26 and 32 wGA between December 2014 and June 2015. These infants were divided into two groups accord- ing to age (26-30 wGA and 30-32 wGA).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
specific temporal TTA-SW | 2 months
  The objective of this study is to evaluate the spatial organization of the specific Temporal theta slow-wave activity (TTA-SW) with the Low-Density Electroencephalography (LD-EEG) at an early stage of development in humans to demonstrate that TTA-SW were independent of auditory stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Wallois, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No